CLINICAL TRIAL: NCT03222479
Title: Development of Stress Guide for Employees: Smartphone-based Stress Management Intervention
Brief Title: Smartphone-based Stress Management Intervention for Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1206/158-112
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Healthy individuals recruited through advertisement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): All individual is instructed to use the application we developed for 4 weeks
  Interventions: Behavioral: Stress guide

INTERVENTIONS:
Behavioral: Stress guide — smartphone-based application that can evaluate stress level and teach how to manage their stress

SUMMARY:
Participants were able to use the application the investigators developed for four weeks. With the application, the participants were able to monitor their stress level and life style patterns. The participants were also provided personalized stress management techniques including psychoeducation and cognitive behavioral technique. In 2014, additional relaxation techniques-abdominal breathing, progressive muscular relaxation, and meditation-were incorporated. Participants' mental health status and life style patterns were evaluated at baseline and at 4 weeks. Pre- and post-intervention statuses were compared after adjusting for degrees of life stress factors. Brief encounter psychosocial instrument (BEPSI-K) score and Center for Epidemiologic Studies Depression Scale (CES-D) score were used as primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Any employee from three corporations (the Korea Gas Corporation (KOGAS), the Korea District Heating Corporation (KDHC), and the Korea Expressway Corporation (KEC)); any individual who visited the health promotion center for a health checkup at Seoul National University Bundang Hospital

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Center for Epidemiologic Studies Depression Scale (CES-D) score at 4 weeks | Baseline and after the intervention for 4 weeks
  Change from baseline Center for Epidemiologic Studies Depression Scale (CES-D) score at 4 weeks
Change from baseline Brief encounter psychosocial instrument (BEPSI-K) score at 4 weeks | Baseline and after the intervention for 4 weeks
  Change from baseline Brief encounter psychosocial instrument (BEPSI-K) score at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hyun Kim, MD, Ph.D, Principal Investigator — Seoul National Univerysity Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No